CLINICAL TRIAL: NCT06702462
Title: A Randomized, Non-inferiority, Double-blind, Controlled, Single-dose, 2-way Cross-over Study to Assess the Potential for Airway Sensitivity Reactions With Propellants HFA-152a (Test) and HFA-134a (Reference) Administered Via Pressurized Metered Dose Inhalers in Adults Aged 18-45 With Mild Asthma
Brief Title: A Study to Assess the Potential for Airway Sensitivity Reactions With Propellants HFA-152a (Test) and HFA-134a (Reference) Administered Via Pressurized Inhalers in Adults With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 223166
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Asthma; HFA-152a; HFA-134a; pMDI
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HFA-152A propellant followed by HFA-134A propellant (Experimental)
  Interventions: Drug: HFA-152A propellant; Drug: HFA-134A propellant
- HFA-134A propellant followed by HFA-152A propellant (Experimental)
  Interventions: Drug: HFA-152A propellant; Drug: HFA-134A propellant

INTERVENTIONS:
Drug: HFA-152A propellant — HFA-152A propellant is administered via oral inhalation
Drug: HFA-134A propellant — HFA-134A propellant is administered via oral inhalation

SUMMARY:
The purpose of the study is to assess the propellants,1 - Difluoroethane [HFA-152a] (Test) and 1,1,1,2-Tetrafluoroethane [HFA-134a] (Reference) for their potential to cause the airways to tighten when delivered through pressurized metered dose inhalers (pMDI). The rationale for this study is to develop a low carbon footprint alternative propellant, HFA-152a, which will have a lower impact on global warming.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study if all the following criteria apply:

* Male or female; females may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
* Participant must be 18 to 45 years of age inclusive, at the time of screening.
* Confirmed diagnosis of asthma: documented, established diagnosis of asthma for at least 6 months.
* Receiving 1 of the following asthma treatments, at a stable dose, for at least 12 weeks prior to the screening visit and is anticipated to remain stable for the duration of the study:

  * As needed short-acting beta-agonists (SABA) only
  * As needed SABA plus low-dose Inhaled corticosteroids (ICS) (defined as 100-250 µg/day fluticasone propionate or equivalent taken whenever SABA is taken).
  * Daily maintenance low-dose ICS, plus as needed SABA or ICS-SABA single inhaler combination therapy
  * Low dose combination single inhaler ICS-formoterol or single inhaler ICS-SABA as needed for symptom relief (and if needed, before exercise)
  * Leukotriene receptor antagonist (LTRAs) in combination with any of the above therapies
* Asthma Control Questionnaire (ACQ)-6 score <1.5 at screening and Day -1.
* No severe asthma exacerbations within 6 months prior to screening and ≤1 severe exacerbation during the 12 months prior to screening.
* Lung function: subjects with a pre-bronchodilator FEV1 ≥60% predicted at Screening and Day-1.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  * Is a Woman of non-childbearing potential (WONCBP) OR
  * Is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of <1%.
* Female participants must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 28 days before the first dose of study intervention.
* For male participants, no contraceptive measures are required.
* Non-smokers, or previous smokers who have not used any tobacco containing-products or vaping products within 12 months prior to study start, and with a total pack year history of ≤10 pack years.
* The use of marijuana, even with a valid prescription, is prohibited within 12 months prior to study start.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* A history of life-threatening asthma or asthma that is unstable in the opinion of the investigator.
* Asthma treatment requiring use of biologic agents (e.g. mepolizumab or dupilumab), chronic systemic corticosteroids, or oral controller agents other than LTRAs.
* Respiratory disorders other than asthma; A history of respiratory diseases to include (but not limited to): pneumothorax, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, cystic fibrosis, bronchiectasis, interstitial lung disease, emphysema, chronic obstructive pulmonary disease, tuberculosis and other respiratory abnormalities other than asthma that, in the opinion of the investigator, would put the participant at risk through study participation, or would affect the study analyses if the disease exacerbates and/or requires additional therapy during the study. This includes history of lung cancer and previous thoracic surgery such as lung resection.
* Asthma Exacerbation: Any severe asthma exacerbation within 6 months prior to screening. (Severe asthma exacerbation defined as a deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days, or a single depo injection or an in-patient hospitalization or early discontinuation (ED) visit due to asthma that required systemic corticosteroids).
* Biologic/immunosuppressive therapies that can be used for the treatment of respiratory diseases during the 6 months, or 5 half-lives whichever is longer-prior to start of the study.
* Participants undergoing de-sensitization therapy.
* Administration of systemic, oral, or depot corticosteroids for asthma treatment within 12 weeks of Visit 1. Intranasal corticosteroids are permitted if at a stable dose for at least 3 months prior to screening.
* Stable doses (3 months or longer) of the following are permitted:

  * Intranasal corticosteroids
  * Oral anti-histamines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Forced expiratory volume in 1 second (FEV1) at 15 minutes | Baseline (0 minutes) and at 15 minutes post dose

SECONDARY OUTCOMES:
Area under the forced expiratory volume in 1 second-time curve from zero to 15 minutes (FEV1 AUC0-15min) | Up to 15 minutes post dose
Percentage change from baseline in FEV1 at 5, 60 and 180 minutes | Baseline (0 minutes) and at 5, 60 and 180 minutes post dose
Percentage change from baseline in FEV1 <-15% at timepoints 5, 15, 60 and 180 minutes | Baseline (0 minutes) and at 5, 15, 60 and 180 minutes post dose
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 54 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf